CLINICAL TRIAL: NCT03991195
Title: Regulatory Mechanism of Intestinal Microorganism in Intervening Mild Cognitive Impairment Based on Multi-modal Neuroimaging Techniques
Brief Title: Intervention of Intestinal Microorganism in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XuanwuH 2 (Other)
Collaborators: First Hospital of Tsinghua University (Other); Beijing Normal University (Other)
Responsible Party: Sponsor-Investigator, XuanwuH 2, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HanYingsc
Record Dates: First submitted 2019-04-28; First posted 2019-06-19 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Gut Microbiota; Mild Cognitive Impairment; Dementia, Alzheimer Type; Neuroimaging
Keywords: mild cognitive impairment; intestinal microorganism; regulation; magnetic resonance imaging
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic supplemented group with aMCI (Experimental): Thirty participants in this group will take Bifidobacterium for three months.
  Interventions: Dietary Supplement: Probiotic supplemented intervention
- Placebo group with aMCI (Placebo Comparator): Thirty participants in this group will take placebo for three months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic supplemented intervention — In this project, taking the method of random, double blindness and control, the probiotic supplemented group with aMCI will take Bifidobacterium for three months. After that, cognitive changes will be test to investigate the effectiveness of probiotic supplementation.
  Arms: Probiotic supplemented group with aMCI
Dietary Supplement: Placebo — In this project, taking the method of random, double blindness and control, the placebo group with aMCI will take placebo for three months. After that, cognitive changes will be test.
  Arms: Placebo group with aMCI

SUMMARY:
Alzheimer's disease (AD) is the most common form of neurodegenerative disorders leading to dementia. Currently, there has been no effective drugs targeting this disease. Dysbiosis of the gut microbiota is considered to be associated with AD, and probiotic supplementation may positively affect cognitive function. However, there are few studies involving the relationship between intestinal microorganism and amnestic mild cognitive impairment (aMCI). In this project, taking the method of random, double blindness and control, the probiotic supplemented group with aMCI will take certain Bifidobacterium for a certain time. After that, the investigators aim to investigate the improvement of cognitive function and changes of intestinal microbial flora diversity via combining neuropsychological tests and 16S recombinant deoxyribonucleic acid (rDNA) high-throughput sequencing technique. Furthermore, based on the multi-modal neuroimaging techniques, the regulatory mechanism of intestinal microorganism in intervening aMCI will be revealed from the perspective of brain networks. In conclusion, these results are beneficial for understanding the therapeutic effect of gut microbiota as a non-drug treatment for early AD and further elucidating the potential brain mechanism, which are of great values in solving scientific and clinical practice issues.

DETAILED DESCRIPTION:
Dysbiosis of the gut microbiota is considered to be associated with Alzheimer's disease (AD), and probiotic supplementation may positively affect cognitive function for patients with AD. However, there are few existing studies involving the role of gut microbiota in possible intervention for amnestic mild cognitive impairment (aMCI).

In this project, taking the method of random, double blindness and control, the probiotic supplemented group with aMCI will take Bifidobacterium for three months. The control group with aMCI will take placebo. After that, the investigators aim to investigate the differences of cognitive function between these two groups and changes of intestinal microbial flora diversity via combining neuropsychological tests and 16S rDNA high-throughput sequencing technique. Furthermore, based on the multi-modal neuroimaging techniques, including structural magnetic resonance imaging (sMRI）, functional MRI, diffusion tensor imaging (DTI)， functional near-infrared spectroscopy (fNIRS), the regulatory mechanism of intestinal microorganism in intervening aMCI will be revealed from the perspective of brain networks.

In conclusion, these results are beneficial for understanding the therapeutic effect of gut microbiome as a non-drug treatment for early AD and further elucidating the potential brain mechanism, which are of great values in solving scientific and clinical practice issues.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of patients with aMCI: memory loss complaint confirmed by an informant; objective cognitive impairment in single or multiple domains, adjusted for age and education; preserved general cognitive function; failure to meet the criteria for dementia; the clinical dementia rating (CDR) score is 0.5.
* Clinical diagnosis of patients with subjective cognitive decline (SCD): presence of self-perceived continuous cognitive decline compared to previous normal status and unrelated to an acute event; failure to meet the following criteria for MCI.
* Clinical diagnosis of the control group: no complaint of memory loss; CDR score is 0; no severe visual or auditory impairment.

Exclusion Criteria:

* a history of stroke;
* major depression (Hamilton Depression Rating Scale score > 24 points);
* other central nervous system diseases that may cause cognitive impairment, such as Parkinson's disease, tumors, encephalitis and epilepsy;
* cognitive impairment caused by traumatic brain injury;
* systemic diseases, such as thyroid dysfunction, syphilis and HIV;
* a history of psychosis or congenital mental growth retardation.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-08-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Improvement of Montreal cognitive assessment (MoCA) | Three months
  After intervention for three months, the investigators first aim to compare cognitive changes of Montreal cognitive assessment (MoCA) among three groups, in order to investigate the therapeutic effectiveness of probiotic supplementation and functional foods.
Improvement of Auditory Verbal Learning Test (AVLT) | Three months
  After intervention for three months, the investigators will then compare cognitive changes of Auditory Verbal Learning Test (AVLT) among three groups, in order to investigate the therapeutic effectiveness of probiotic supplementation and functional foods.
Changes of intestinal microbial flora diversity | Three months
  After intervention for three months, the investigators will further compare the diversity changes of intestinal microbial flora, such as Lactobacteria species, Bifidobacterium, Enterococci, Propionobacteria, Peptostreptococci, etc., among three groups.

SECONDARY OUTCOMES:
Structural MRI-based brain network changes | Three months
  After intervention for three months, the investigators will compare the structural changes of brain network among three groups (e.g., efficiency, clustering, modularity) in order to reveal the regulatory mechanism of intestinal microorganism in intervening aMCI.
Functional MRI-based brain network changes | Three months
  After intervention for three months, the investigators will compare the functional changes of brain network among three groups (e.g., functional connectivity, hub) in order to reveal the regulatory mechanism of intestinal microorganism in intervening aMCI.
FNIRS-based brain network changes | Three months
  After intervention for three months, the investigators will compare the functional changes of brain network among three groups (e.g., functional connectivity, small word, efficiency) in order to reveal the regulatory mechanism of intestinal microorganism in intervening aMCI.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, PhD, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- Department of Neurolgy, Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The information of neuropsychological tests, neuroimaging data are to be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: When summary data are published or starting 6 months after publication.
Access Criteria: The information of neuropsychological tests, neuroimaging data will be shared.